CLINICAL TRIAL: NCT01554709
Title: A Study to Collect Additional Information Related to the Safety and Performance of the CardioGard Cannula
Brief Title: Safety and Performance Study of the CardioGard Cannula
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CardioGard Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN0009
Record Dates: First submitted 2012-03-11; First posted 2012-03-15 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Aortic Valve Replacement
Keywords: bypass; cannula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CardioGard Cannula (Experimental)
  Interventions: Device: Aortic Cannulas (CardioGard)
- Reference Cannula (Active Comparator)
  Interventions: Device: Aortic Cannulas (CardioGard)

INTERVENTIONS:
Device: Aortic Cannulas (CardioGard) — Comparison of aortic cannulas during by pass surgery

SUMMARY:
The objective of the study is to collect additional information related to the safety and performance of the CardioGard Cannula during bypass procedures.

ELIGIBILITY:
Inclusion Criteria:

* AVR (Aortic Valve Replacement), AVR+CABG (Coronary Artery Bypass Surgery)
* Non pregnant female

Exclusion Criteria:

* Contraindication for open heart surgery under bypass machine
* Emergency Operation

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
DWI- Diffusion Weighted Imaging | The outcome measure is assessed in average a week after the surgery
  diffusion weighted magnetic resonance imaging (DW-MRI)

SECONDARY OUTCOMES:
TCD- Transcranial Doppler | The Outcome measure is assessed during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gil Bolotin, Dr., Principal Investigator — Rambam Health Care Campus
Locations (5):
- Germany (2):
  - Kerckhoff Klinik, Bad Nauheim
  - Heart Center Leipzig, University of Leipzig, Leipzig
- Rambam Health Care Campus, Haifa, Israel
- Switzerland (2):
  - Insel Hospital, Bern
  - University Hospital Zurich, Zurich